CLINICAL TRIAL: NCT04728880
Title: Remdesivir in Adults With Covid-19: Mansoura University Hospital Experience
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mostafa Bakeer, Lecturer of chest medicine, Mansoura University
Other Study IDs: R.20.11.1097
Record Dates: First submitted 2021-01-26; First posted 2021-01-28 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2021-01

CONDITIONS: Pneumonia, Viral
MeSH Terms: conditions — Pneumonia, Viral | interventions — remdesivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Remdesivir — This study is a retrospective trial to assess the efficacy of Remdesivir in adult patients diagnosed with COVID-19 in Mansoura University Isolation Hospital. In this study we will analyze the data collected during treatment.

SUMMARY:
COVID-19 is a respiratory disease caused by a new coronavirus (SARS-CoV-2) and causes significant morbidity and mortality. This study is a retrospective trial to assess the efficacy of Remdesivir in adult patients diagnosed with COVID-19 in Mansoura University Isolation Hospital. In this study the investigators will analyze the data collected during treatment.

DETAILED DESCRIPTION:
COVID-19 is a novel respiratory disease caused by coronavirus (SARS-CoV-2) and results in significant morbidity and mortality. To date there is no approved medication for the treatment of patients with COVID-19. Remdesivir is a broad-spectrum antiviral nucleotide analogue that inhibits RNA-dependent RNA polymerase activity among a diverse group of RNA viruses. Non-clinical and clinical data suggest that Remdesivir may be useful for the treatment of COVID-19. WHO has identified Remdesivir as a candidate drug of interest to be studied in clinical trials. This retrospective study is designed to analyze the data collected during the routine care of patients who have benefited from this therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 18 years old.
2. SARS-CoV-2 infection confirmed.
3. Patients having classical radiological lesions of COVID-19 on X-ray chest or HRCT chest.
4. Hospitalized patients who received at least one administration of Remdesivir therapy (Dose: 200mg day one then 100mg daily for up to 10 days).

Exclusion Criteria:

1. Presences of chronic renal failure > 4 stage, GFR < 30ml/min.
2. ALT/AST > 5 times than normal values.
3. Pregnant women.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with COVID-19 in Mansoura University Isolation Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-26 (Estimated); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-05-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Pulse rate | 15 days
  Change from baseline in the pulse rate during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in respiratory rate | 15 days
  Change from baseline in the respiratory rate during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in body core temperature | 15 days
  Change from baseline in the body core temperature during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in blood pressure | 15 days
  Change from baseline in the blood pressure during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in arterial blood gas analyses | 15 days
  Change from baseline in the arterial blood gas analyses during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in Spo2 / FIO2 ratio | 15 days
  Change from baseline in the Spo2 / FIO2 ratio during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in White blood cell count | 15 days
  Change from baseline in the White blood cell count during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in lymphocyte count | 15 days
  Change from baseline in the lymphocyte count during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in lactate dehydrogenase | 15 days
  Change from baseline in the lactate dehydrogenase during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in D-dimer | 15 days
  Change from baseline in the D-dimer during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in procalcitonin | 15 days
  Change from baseline in the procalcitonin during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in Interleukin-6 | 15 days
  Change from baseline in the Interleukin-6 during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in Serum ferretin | 15 days
  Change from baseline in the Serum ferretin during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in prothrombin time | 15 days
  Change from baseline in the prothrombin time during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in serum creatinine | 15 days
  Change from baseline in the serum creatinine during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in liver enzyme ALT | 15 days
  Change from baseline in the liver enzyme ALT during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in creatinine kinase | 15 days
  Change from baseline in the creatinine kinase during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in cardiac troponin | 15 days
  Change from baseline in the cardiac troponin during clinical course of patients on Day 15 under treatment with Remdesivir.
Change from baseline in The Sequential Organ Failure Assessment score (SOFA score) | 15 days
  The Sequential Organ Failure Assessment (SOFA) is a morbidity severity score and mortality estimation tool. It allows for calculation of both the number and the severity of organ dysfunction in six organ systems (respiratory, coagulatory, liver, cardiovascular, renal, and neurologic). The following values are used to calculate the score: (PaO2 / FiO2 and artificial ventilation; platelets; bilirubin; average blood pressure and use of vasoactive drugs; creatinine).The total score ranges from 0-24. Zero indicates low risk while 24 indicates higher risk of mortality.

SECONDARY OUTCOMES:
Duration of hospitalization | 15 days
  Number of days of hospital admission either in ICU or ward till date of discharge
Supplemental Oxygen Requirement from Baseline | 15 days
  Duration of increased supplemental oxygen requirement from baseline
Duration without mechanical ventilation | 15 days
  Duration without mechanical ventilation within 15 days of initiation of treatment with Remdesivir
Mortality | 15 days
  Mortality at 15 days after initiation of treatment with Remdesivir.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Hospital, Al Mansurah, Dakahliya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided